CLINICAL TRIAL: NCT00517348
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IMA-026 Administered Subcutaneously or Intravenously to Healthy Subjects
Brief Title: Study Evaluating IMA-026 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3192K1-1000
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Adult

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: IMA-026 — SC and IV ascending single doses from lyophilized dosage form 0.3, 1, 2, 4 mg/kg SC and 3 mg/kg IV

SUMMARY:
To assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of IMA-026 administered subcutaneously (SC) or intravenously (IV) in healthy adults.

ELIGIBILITY:
* Healthy men and women ages 18 - 50
* Body weight greater than or equal to 50 kilograms
* Nonsmoker or fewer than 10 cigarettes per day
* No serious infection, i.e., requiring hospitalization or IV antibiotics, or an upper respiratory infection within 1 month before dosing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) analysis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- San Antonio, Texas, United States